CLINICAL TRIAL: NCT05710458
Title: Performance Comparison of the 25 Gauge 20,000cpm HYPERVIT Dual Blade vs. 10,000cpm ULTRAVIT Vitrectomy Cutter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Nicholas Fung, Clinical Asst Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20K
Record Dates: First submitted 2023-01-25; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Vitrectomy; Epiretinal Membrane; Macular Hole; Vitreous Hemorrhage; Retinal Detachment
MeSH Terms: conditions — Epiretinal Membrane; Retinal Perforations; Vitreous Hemorrhage; Retinal Detachment

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients are randomised and masked from the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25 gauge 20,000 cpm Hypervit Dual Blade (Experimental): New vitrectomy blade with higher cutting rate
  Interventions: Device: 25 gauge 20,000 cpm Hypervit Dual Blade
- 25 gauge 10,000 Ultravit vitrectomy cutter (Active Comparator): Existing vitrectomy blade with cutting rate 10,000 cut/min
  Interventions: Device: 25 gauge 10,000 cpm Ultravit Vitrectomy Cutter

INTERVENTIONS:
Device: 25 gauge 20,000 cpm Hypervit Dual Blade — Vitrectomy blade with increased cutting rate to 20,000 cut/min
  Other Names: 20K
  Arms: 25 gauge 20,000 cpm Hypervit Dual Blade
Device: 25 gauge 10,000 cpm Ultravit Vitrectomy Cutter — Existing Vitrectomy blade with cutting rate 10,000 cut/min
  Other Names: 10K
  Arms: 25 gauge 10,000 Ultravit vitrectomy cutter

SUMMARY:
This prospective randomised controlled trial will be conducted to investigate that increasing the vitrectomy cutting rate from 10,000 cut/min to 20,000 cut/min will result more efficiency and shorter core vitrectomy time, and it is equally safe as compared to the current 10,000 cut/min. We plan to target the patients undergoing for vitrectomy for common vitreoretinal pathology. Our plan is to conduct a randomised study with 2 arms, one with the higher cutting rate (20,000 cut/min) versus a second arm using the existing system 10,000 cuts/min.

DETAILED DESCRIPTION:
In addition, we will measure the core vitrectomy duration by Constellation Vision System stopwatch. We will count the duration when the vitrectomy probe enter into the eye to the moment the performing the air/fluid exchange by shaving the peripheral vitreous to complete the vitrectomy. For our second outcome measure to prove the no-inferiority of intraoperative and postoperative complications patients will have 3 months follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age who are undergoing vitrectomy for the following conditions:

  * Macular hole
  * Epimacular membrane
  * Vitreous hemorrhage
  * Primary retinal detachment

Exclusion Criteria:

* Patient who is

  * unable to give proper consent
  * previous vitrectomy or scleral buckle surgery
  * cases requiring silicone oil tamponed
  * undergoing repeated retinal detachment surgery
  * undergoing surgery for tractional diabetic retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Duration of Core vitrectomy | intraoperative (From the moment probe enter into the eye till performing the air/fluid exchange to complete the vitrectomy)
  Measurement of core vitrectomy duration by Constellation Vision System

SECONDARY OUTCOMES:
Non-inferiority of intraoperative and postoperative complication | 3 months
  Safety and Efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Grantham Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
By direct contact to the corresponding author or PI
Supporting Information: Study Protocol, CSR
Time Frame: 5 Years after the study ends
Access Criteria: Case by case

REFERENCES:
- [Background] O'Malley C, Heintz RM Sr. Vitrectomy with an alternative instrument system. Ann Ophthalmol. 1975 Apr;7(4):585-8, 591-4. PMID 1147502
- [Background] Rizzo S, Genovesi-Ebert F, Belting C. Comparative study between a standard 25-gauge vitrectomy system and a new ultrahigh-speed 25-gauge system with duty cycle control in the treatment of various vitreoretinal diseases. Retina. 2011 Nov;31(10):2007-13. doi: 10.1097/IAE.0b013e318213623a. PMID 21685823